CLINICAL TRIAL: NCT04852809
Title: The Utilisation of Technology and Its Impact on Clinical Trial Patient Care During the Coronavirus Pandemic 2020-2021
Brief Title: COvid-19 aNd TechNology - thE Impact on Clinical Trial Patients
Acronym: CONNECT
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp197
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Questionnaire: Observational
  Interventions: Other: No intervention
- Focus Group: Observational
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
This is a 2 part qualitative study involving a questionnaire (part 1) and focus group discussions (part 2).

The purpose of the study is to evaluate how patients' attitudes to technology in the oncology clinical trials setting since the start of the Coronavirus pandemic in 2020, and to assess how their use of technology has changed during this time.

Part 1 of the study will be conducted via a self-report questionnaire to 100-140 cancer patients involved in clinical trials at The Christie NHS Foundation Trust over a 2 month period. Following this, three focus groups with a maximum of 8 participants in each group will take place to further assess patients' experiences with technology during the pandemic.

Participants may take part in part 1 or part 2 only, or in both.

DETAILED DESCRIPTION:
Clinical trial involvement is more resource-intensive than receiving standard of care treatment and often results in more frequent hospital visits for patients. To reduce the risk of patients to COVID-19, there has been a shift towards reducing on-site visits with increased use of technology e.g. virtual visits. Patients may have also been using devices at home to aid in their care, including digital devices, mobile applications, smart watches and, rarely, trial-specific devices, to monitor aspects of their own health.

Our project will explore the impact that the coronavirus pandemic has had on clinical trial patients and how they feel technology could help or create barriers in their future care.

In order to quantify how clinical trial visits have changed and to evaluate patient's attitudes to the increasing use of technology in clinical trials, we will be disseminating questionnaires to 100 patients currently on clinical trials over a 2 month period. We will follow these up with three virtual focus group discussions with 8 participants in each to delve further into patients' experiences.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Patients have to be 18 years of age or older.
2. Patients have to be currently enrolled on a phase I, II or III cancer related clinical trial within the Christie NHS Foundation Trust

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Unable to understand and converse in English for the focus group session.
2. Patient not currently involved in a phase I, II or III clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will all be clinical trial patients from The Christie NHS Foundation Trust who meet the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
To evaluate patients' attitudes to technology in the clinical trial setting since the coronavirus pandemic 2020. | 9 months

SECONDARY OUTCOMES:
To assess changes in patients use of technology in oncology clinical trials prior to and since the coronavirus pandemic 2020. | 9 months

OTHER OUTCOMES:
To determine how coronavirus pandemic has impacted the use of technology in the delivery of oncology trials for patients. | 9 months
To assess the relationship between socioeconomic status and age and how it impacts the use of technology | 9 months
To evaluate the challenges and opportunities of using technology in the future in the delivery of clinical trials technologies for future patient care. | 9 months
To assess the role of healthcare technologies for future patient care. | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HRA website for results summary — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/